CLINICAL TRIAL: NCT05738811
Title: Effectiveness of EMS Versus TENS During Gait Training in Post Stroke Patients to Improve Gait and Quality of Life A Randomized Clinical Trial
Brief Title: Effectiveness of EMS Versus TENS During Gait Training in Post Stroke Patients to Improve Gait and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Principal Investigator, Waseem Javaid, Project Director, Sehat Medical Complex
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zunairaahmad23
Record Dates: First submitted 2023-02-11; First posted 2023-02-22 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Stroke, Anterior Cerebral Artery
MeSH Terms: conditions — Infarction, Anterior Cerebral Artery | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS treatment group (Experimental): Group A was given exercise protocol along with TENS treatment protocol.
  Interventions: Other: TENS treatment protocol; Other: Exercises
- EMS treatment group (Experimental): Group B received exercise protocol along with EMS treatment protocol.
  Interventions: Other: EMS treatment protocol; Other: Exercises

INTERVENTIONS:
Other: TENS treatment protocol — The 2 sets of electrodes of TENS were placed over the common peroneal nerve as it passes over the head of fibula and the motor point of tibialis anterior to elicit dorsiflexion and eversion of foot.
  Arms: TENS treatment group
Other: EMS treatment protocol — The electrodes were placed over the common peroneal nerve as it passes over the head of fibula and the motor point of tibialis anterior to elicit dorsiflexion and eversion of foot. A portable comfy EMS channel was used to apply EMS protocol to set at threshold of muscle contraction level.
  Arms: EMS treatment group
Other: Exercises — Patient were given 30 minutes treatment session, 10 minutes of supported walking 10 minutes of BWS treadmill training 10 minutes of Task-specific over ground locomotor training (LT) There was rest of 2 minutes The frequency of the sessions was five times a week for 12 weeks.

SUMMARY:
The goal of this Randomized clinical trial was to compare effectiveness of EMS versus TENS during gait training in stroke patients to improve gait and quality of life. The main question it aims to answer was:

• To compare effectiveness of EMS versus TENS during gait training in post stroke survivors to improve gait and quality of life Participants were given consent form and after subjects read and sign the informed consent, they were included in study according to eligibility criteria. 2 groups were included in study, one group received stimulation through TENS and other through EMS. Both groups received exercise protocol and stimulation would be provided only during gait training. Outcome was measured through different outcome measure tools.

DETAILED DESCRIPTION:
Patients with stroke experience gait disorders due to various causes, including sensory impairment and muscle weakness, spasticity, etc., and the primary goal of rehabilitation is to regain independent walking. The ankle plantar flexors tightly contract to maintain a standing posture and contribute to postural control through anticipatory contractions before changes in the center of mass. The plantar flexors in the ankle create most of the energy required for forward propulsion of body mass during walking. The strength of the ankle plantar flexors on the paretic side is related to the gait speed of patients with stroke. The peripheral sensory inputs via Electrical muscle stimulation enhanced the activities of circuits in the somatosensory cortex thus it can cause neuroplasticity to brain. Electrical stimulation on ankle dorsiflexors could be an effective management to enhance gait performance and ankle control during walking in chronic stroke patients. Neuromuscular electrical stimulation on ankle plantar flexors may improve gait symmetry. When neuromuscular stimulation combined with activity can enhance efficacy. Many previous studies conducted trials on effectiveness of muscle stimulation but this study aims to perform a clinical trial to enhance evidence about effectiveness.

2 groups were included in study, one group received stimulation through TENS and other through EMS. Both groups received exercise protocol and stimulation was provided only during gait training. The outcome was measured through different outcome measure tools.

Functional electrical stimulation device was used to improve dorsiflexion during walking, but it was somehow expensive treatment. To achieve same outcome during walking, it is aimed to see effect of EMS vs TENS. This would be an inexpensive alternate of FES device and could improve gait and quality of life if used during treatment protocol. So it was aimed to generate evidence about effectiveness of TENS vs EMS on lower limb during gait training to improve gait and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subacute Stroke Patients referred from neurophysician
* Anterior cerebral artery lesion
* Age between 40-70 years
* Well-oriented patients (ability to understand and follow simple verbal instructions)
* Ambulatory before stroke
* Ability to stand with or without assistance and to walk at least 10 meter with or without assistance

Exclusion Criteria:

* Red flags to walking or to electric stimulation
* History of peroneal nerve lesions
* Cognitive impairment
* Fixed plantar-flexor contractures
* Knee deformity

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-02-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Wisconsin gait scale (change is being assessed) | Change from Baseline at 12 weeks
  Wisconsin Gait Scale is an observational tool for the evaluation of gait quality in individuals after stroke with hemiplegia. It is divided into four subscales, which assess a total of fourteen spatiotemporal and kinematic parameters of gait observed during the consecutive gait phases.
  Minimum score is 13.35, highest the score, the more the gait is affected.
10 meter walk test (change is being assessed) | Change from Baseline at 12 weeks
  The individual is instructed to walk a set distance (6 meters, 10 meters, etc). Time is measured while the individual walks the set distance (often the individual is given space to accelerate to his/her preferred walking speed (this distance is not included when determining speed).
Stroke specific quality of life scale (change is being assessed) | Change from Baseline at 12 weeks
  Specific Quality Of Life scale is a patient-centered outcome measure intended to provide an assessment of health-related quality of life specific to patients with stroke. Scores range from 49-245. Higher scores indicate better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Zunaira Ahmad, Principal Investigator — University of Lahore
Locations (1):
- Sehat Medical Complex, Lahore, Lahore, Punjab Province, Pakistan